CLINICAL TRIAL: NCT00474474
Title: Study of the Impact of How the Virtual Patient's Anamnesis is Designed on the Reasoning Pattern and Therapeutic Decision Making
Brief Title: Study of the Impact of Virtual Patient Designs on the Reasoning Pattern and Therapeutic Decision Making
Acronym: VPtdl-rct1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: VP-02-001
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Decision Making; Computer-Assisted
Keywords: virtual patient; therapeutic decision making

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Virtual patient is NOT introduced

SUMMARY:
There is a lack of evidence of the impact of the information provided in the introduction screen on the students diagnostic and therapeutic decisions. The reasoning pattern may also be altered if positive findings are provided to the student without an active request for it.

The results will be of importance when virtual patients are used for assessing students.

DETAILED DESCRIPTION:
The problem-solving approach is found in virtual patient designs concerned with teaching clinical reasoning and diagnosis. Generally the student has to collect a range of information, usually from menus of possible history questions, physical examination, and lab tests, and make diagnostic and therapeutic decisions based on their findings. The information is not cued - the student have to decide what is relevant. An introduction screen is shown to the student when the virtual patient is initiated. Case author have used it differently - some entered a complete chief complaint and part of anamnesis findings while other have not disclosed anything about the patient. There is a lack of evidence of the impact of the information provided in the introduction screen on the students diagnostic and therapeutic decisions. The reasoning pattern may also be altered if positive findings are provided to the student without an active request for it.

The results will be of importance when virtual patients are used for assessing students.

ELIGIBILITY:
Inclusion Criteria:

* All the students enrolled in the comprehensive dentistry course at the time of the study (2007)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
therapeutic decision making | 1 hour

SECONDARY OUTCOMES:
Medical history reasoning (required/unnecessary) | 1 hour
Time allocation to the different phases in solving a VP | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Uno Fors, Principal Investigator — LIME, Karolinska Institutet
Locations (1):
- School of dentistry, Karolinska Institutet, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Zary N, Johnson G, Boberg J, Fors UG. Development, implementation and pilot evaluation of a Web-based Virtual Patient Case Simulation environment--Web-SP. BMC Med Educ. 2006 Feb 21;6:10. doi: 10.1186/1472-6920-6-10. PMID 16504041